CLINICAL TRIAL: NCT00871819
Title: Optimized Programming in a Multiple-Independent Current Sources Spinal Cord Stimulation (SCS) System
Brief Title: Optimized Programming in Spinal Cord Stimulation (SCS) System
Acronym: OP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: A2008
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Neuropathic Pain; Pain
Keywords: Spinal Cord Stimulation
MeSH Terms: conditions — Neuralgia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal Cord Stimulation Group (Other): Spinal Cord Stimulation (SCS) Treatment Group
  Interventions: Device: Precision Spinal Cord Stimulation (SCS)

INTERVENTIONS:
Device: Precision Spinal Cord Stimulation (SCS) — Various SCS device programming parameters
  Other Names: Precision Spinal Cord Stimulation System

SUMMARY:
The objective of this study is to evaluate extent, location, and perception of paresthesia as a function of anode/cathode configuration.

DETAILED DESCRIPTION:
The clinical results from this study may help to validate predictions made by mathematical models of neurons that are activated by SCS and increase scientific knowledge about the way in which different programs relate to satisfactory outcomes, such that use of the model may help in the development of new products.

ELIGIBILITY:
Inclusion Criteria:

* Be previously implanted with Precision SCS System (3-36 months post permanent implant) having 2 parallel percutaneous leads placed between T8-T10.
* Be implanted with Precision SCS System for the treatment of neuropathic pain of trunk and/or limbs
* Be 18 years of age or older
* Be extremely satisfied, very satisfied, or satisfied with SCS therapy for treatment of pain condition
* Be able to use pen tablet to document regions of paresthesia and pain
* Be able to lie in the supine position for 45 minutes at a minimum
* Be able to verbally report qualitative and quantitative aspects of paresthesia sensations.
* Have a paresthesia threshold on a standard program below 4mA while in the supine position
* Have at minimum the upper contact of one lead below T8 and the lower contact above T11 vertebral levels
* Be willing and able to comply with study-related procedure
* Agree to study requirements and provides written Informed Consent

Exclusion Criteria:

* Unable to read, write, speak, and understand English
* Currently pregnant or planning to become pregnant during the course of the study
* Have negative finding in any of the pre-screening and screening requirements
* Upon fluoroscopy, location of both leads is identified to be outside T8-T10 vertebral levels
* Unable to perceive the sensation of paresthesia associated with stimulation in the trunk and/or lower extremities
* Have a drug pump and/or a non-Precision neurostimulation device (regardless of whether active or inactive)
* Have had any interventional pain procedure or surgeries (including Interlaminar epidural steroid injection, Transforaminal epidural steroid injection, Caudal epidural steroid injection, Selective nerve root block, Intraarticular lumbar facet injection, Sacroiliac joint injection, Piriformis muscle injection, Trochanteric bursa injection, Hip/knee joint injections, Medial branch block (innervates facet joint), Pulsed radiofrequency neurotomy medial branches, Pulsed radiofrequency dorsal root ganglion, Thermal (high temperature) radiofrequency neurotomy medial branches, Trigger point injections, and Botulinum toxin injections) involving the spine within the past 30 days
* Have any condition that is likely to confound evaluation of study endpoints. Conditions that may make paresthesia coverage variable over the course of the study include multiple sclerosis, partial spinal cord injury, diabetic peripheral neuropathy, peripheral vascular disease, scoliosis, deafferentation, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Kormylo, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spinal Cord Stimulation Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Stimulation Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient Between Dorsal Root Paresthesia (Total Pixels Derived From Digital Drawing) at Maximum-comfortable Stimulation Level and Anode-cathode Separation Distance (mm)
Time Frame: Immediately post-procedure
Measure: Number; unit: Correlation coefficient
Groups:
- All Subjects: All enrolled subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Correlation coefficient | 0.6202

ADVERSE EVENTS:
Arm/Group | Spinal Cord Stimulation Group
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Small number of subjects; technical outcomes not necessarily predictive of therapeutic effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less